CLINICAL TRIAL: NCT00380497
Title: Pico-Salax Versus Poly-Ethylene Glycol for Bowel Cleanout Before Colonoscopy in children-a Single Blinded Randomized Controlled Trial
Brief Title: Pico-Salax Versus Poly-Ethylene Glycol for Bowel Cleanout Before Colonoscopy in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Simon Ling, Staff Gastroenterologist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1000008846
Record Dates: First submitted 2006-09-25; First posted 2006-09-26 (Estimated); Last update posted 2013-07-29 (Estimated); Status verified 2013-07

CONDITIONS: Colonoscopy
Keywords: Pediatrics; Colonoscopy; Bowel cleanout; Poly-Ethylene Glycol; Pico-Salax
MeSH Terms: interventions — Pico-Salax

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pico-Salax (Experimental)
  Interventions: Drug: Pico-Salax®
- PEGlyte (Active Comparator)
  Interventions: Drug: PEG-Lyte®

INTERVENTIONS:
Drug: PEG-Lyte®
  Arms: PEGlyte
Drug: Pico-Salax®
  Arms: Pico-Salax

SUMMARY:
The purpose of this trial is to compare patient's satisfaction from Pico-Salax with the standard of care, Poly-Ethylene Glycol and electrolyte solution, for bowel cleanout before colonoscopy in children, and to compare effectiveness.

DETAILED DESCRIPTION:
Good bowel cleanout before colonoscopy is commonly associated with significant discomfort that children do not tolerate well. Many pediatric centers in North America use Poly-Ethylene Glycol and electrolyte solution (PEG-ELS, Golytely®) for bowel lavage administered in a large volume, often causing nausea, vomiting and bloating. This is often poorly tolerated by children who usually require the insertion of a nasogastric tube and a day admission. Recently, Pico-Salax was approved in Canada for bowel cleanout in children. It is administered in two divided doses, each in one cup of water; it is palatable and does not have to be given in hospital. However, no controlled study in children compared it with the current standard of care. Our preliminary experience and previous literature suggest that it is effective and well tolerated. We propose to study whether colon cleanout for colonoscopy with Pico-Salax is better tolerated than Golytely in children, by a single blinded randomized controlled trial. Positive results of this study will facilitate a better tolerated regimen for bowel clean out in children.

ELIGIBILITY:
Inclusion Criteria:

* Children between 4 and 18 years of age
* Undergoing full elective ambulatory colonoscopy

Exclusion Criteria:

* Evidence of bowel obstruction, prior partial or total colectomy and significant renal failure (GFR<50 mls/min/1.73 m2)
* Second dose of Pico-Salax will not be given to children with blood pressure less than the tenth percentile or pulse rate >90th% of normal reference value for age, or in children with a clinical need for bolus IV fluids decided by the clinical fellow

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 83 (Actual)
Dates: Start 2006-09; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Patient's satisfaction from the regimen as assessed by a questionnaire completed by the child and parents

SECONDARY OUTCOMES:
Cleanout effectiveness (measured by: rating of a blinded gastroenterologist, the need for enema supplement, procedure length and whether the planned destination was reached
Side effects (measured by: dehydration assessment, questionnaires completed by the nurse and the patient, and blood tests)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Ling, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada